CLINICAL TRIAL: NCT06686433
Title: Assessing the Impact of a Novel Infant Formula on Immunity, Gut Health and Safety: A Multicenter, Double-blind, Randomized, Controlled Trial
Brief Title: The Impact of a Novel Infant Formula on Immunity, Gut Health and Growth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biostime (Guangzhou) Health Products Limited (Industry)
Collaborators: Merieux NutriSciences (China) (Unknown); BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Pistar2RCT
Record Dates: First submitted 2024-11-10; First posted 2024-11-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy Term Infant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test (Experimental): Novel infant formula
  Interventions: Other: Novel infant formula
- Control (Active Comparator): Standard infant formula
  Interventions: Other: Standard infant formula
- Reference (No Intervention): Breastfeeding

INTERVENTIONS:
Other: Novel infant formula — Infants are fed with the novel infant formula from the date of enrollment to the age of 6 months.
  Arms: Test
Other: Standard infant formula — Infants are fed with the standard infant formula from the date of enrollment to the age of 6 months.
  Arms: Control

SUMMARY:
The goal of this multicenter, double-blind, randomized, controlled trial is to assess the safety and efficacy of a new infant formula on healthy term infants from enrollment to the age of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. At enrollment visit, post-natal age ≤ 42 days (date of birth = day 0).
2. Healthy term infant (≥ 37 weeks of gestation).
3. Infants birth weight ≥ 2500 and ≤ 4500 g.
4. For formula fed group: infant is mainly consuming IF (more than 75% of the infant diet) until at least 4 months of age. The parents / LAR(s) have independently decided NOT to breastfeed.
5. For the breastfed reference group: infant has been mainly consuming breastmilk since birth (more than 75% of the infant diet), and the parents / LAR(s) have made the decision to continue breastfeeding until at least 4 months of age.
6. Evidence of personally signed and dated informed consent indicating that the infant's both parents/LAR(s), as per local regulation, have been informed of all pertinent aspects of the study.
7. Parents/LAR(s) of infants demonstrate willingness and capability to adhere to scheduled visits, fulfill the study protocol requirements, and remain accessible by phone throughout the study duration.

Exclusion Criteria:

1. Conditions requiring infant feedings other than those specified in the protocol.
2. Medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   1. Evidence of major congenital malformation (e.g., cleft palate, extremity malformation)
   2. Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis)
   3. Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigators, would make the infants inappropriate for entry into the study. Of note, infants who are generally healthy but experiencing minor acute illnesses at the time of enrollment, which are common in infancy and do not necessitate any of the exclusionary medications mentioned below, may still be eligible for enrollment.
3. Presently receiving or having received prior to enrolment any medication(s) or supplement(s) which are known or suspected to affect the following:

   1. Fat digestion, absorption, and/or metabolism (e.g. pancreatic enzymes);
   2. Stools characteristics and gut microbiota (e.g., oral, or systemic antibiotics, glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose);
   3. Growth (e.g., insulin or growth hormone);
   4. Gastric acid secretion.
4. Currently participating or having participated in another interventional clinical trial since birth.

Max Age: 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 342 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Daily body weight gain between V1 and V3 | From baseline to the age of 6 months
Fecal total pathogens load | From baseline to the age of 6 months

SECONDARY OUTCOMES:
Secretory IgA, calprotectin and antitrypsin A1 in feces at V1, V2 and V3 | From baseline to the age of 3 months and the age of 6 months
sIgA in saliva at V1, V2 and V3 | From baseline to the age of 3 months and the age of 6 months
Incidence of allergic disease reported by caregivers | From baseline to the age of 3 months and the age of 6 months
Incidence of infectious disease reported by caregivers | from baseline to the age of 3 months and the age of 6 months
Incidence of medications use reported by caregivers | From baseline to the age of 3 months and the age of 6 months
Additional anthropometric measures (body length and head circumference) | From baseline to the age of 3 months and the age of 6 months
GI symptoms and GI-related behaviors assessed via Infant Gastrointestinal Symptom Questionnaire (IGSQ) | From baseline to the age of 3 months and the age of 6 months
Stooling patterns assessed via Amsterdam Infant Stool Scale (AISS) | From baseline to the age of 3 months and the age of 6 months
Overall composition of the fecal microbiota | From baseline to the age of 3 months and the age of 6 months
Fecal metabolome profiles | From baseline to the age of 3 months and the age of 6 months

OTHER OUTCOMES:
The breast milk composition | At baseline only

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Hospital of Southern Medical University, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No